CLINICAL TRIAL: NCT00814216
Title: Randomized, Double-blind, Two Way Cross-over, Proof of Concept Study to Compare Efficacy, Safety, Pharmacokinetics & Pharmacodynamics of QAV680 Versus Placebo, With an Extended Open-label Corticosteroid Period, in Steroid-free, Mild to Moderate Persistent Asthma Patients.
Brief Title: Efficacy, Safety and Pharmacokinetics of QAV680 in Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAV680A2201; EudraCT number: 2008-005168-15
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Efficacy; safety; QAV680; pharmacokinetics; corticosteroid; asthma
MeSH Terms: conditions — Asthma | interventions — NVP-QAV680; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- QAV680 (Experimental)
  Interventions: Drug: QAV680
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo for QAV680
- Fluticasone Propionate Inhaler (Active Comparator)
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: QAV680
  Arms: QAV680
Drug: Matching placebo for QAV680
  Arms: Placebo
Drug: Fluticasone Propionate
  Arms: Fluticasone Propionate Inhaler

SUMMARY:
This study aims to study the efficacy (as measured by change in FEV1) and safety of two-week administration of oral QAV680 in the treatment of patients with asthma.'

ELIGIBILITY:
Inclusion criteria:

* Mild to moderate persistent asthma for at least 6 months.

Exclusion criteria:

* Past or recent history of significant medical illness and/or lab abnormalities including but not limited to ECG abnormalities, abnormal LFT, HIV, Hep B/C,
* Allergic disorders, pancreatic disease, serious underlying respiratory diseases, life threatening asthma, renal disease etc
* Surgical and/or medical conditions which significantly effect ADME of the drug.
* Prior use of asthma medications (except SABA's) prior to 2 weeks of dosing

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Measure: Change in Forced Expiratory Volume in one second (FEV1) as measured by Spirometry. | 2 weeks

SECONDARY OUTCOMES:
Measure: Change in Asthma Control Questionnaire (ACQ) score | 2 weeks
Measure: Frequency of salbutamol usage | 2 weeks
Measure: Change in exhaled Nitric Oxide (NO) | 2 weeks
Home Monitoring Of FEV1 By PIKO Monitors | Day 2 to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, Wiesbaden
- India (4):
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Mysore
  - Novartis Investigative SIte, Nagpur